CLINICAL TRIAL: NCT06795230
Title: Effects of a Low-intensity Muscle Strengthening Protocol in Combination With Blood Flow Restriction Training on Upper Limb Impairment in People With Multiple Sclerosis. A Randomized Controlled Trial
Brief Title: Blood Flow Restriction for Upper Limb Rehabilitation in People With Multiple Sclerosis. A Randomized Controlled Trial (BFRT-EM)
Acronym: BFRT-EM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, Roberto Cano de la Cuerda, PT, PhD. Full Professor, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: UniversidadRJC1
Record Dates: First submitted 2025-01-14; First posted 2025-01-28 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; Upper limb; Rehabilitation; Blood Flow Restriction Training
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: Rehabilitation treatment. We do not use drugs or vaccines.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional muscle strengthening (Active Comparator): Palmar flexion and dorsal flexion; ulnar deviation and radial deviation; pronation and supination; elbow flexion and extension, with a dumbbell at 70% of the 1RM, performing a total of 4 series of 8 - 12 repetitions each, avoiding reaching muscle failure in each series.
  Interventions: Other: Conventional physical therapy
- BFRT (Experimental): The experimental group will carry out a low-intensity strengthening program (20% 1RM) in combination with the BFRT system composed of the following exercises: palmar flexion and dorsal flexion; ulnar deviation and radial deviation; pronation and supination; elbow flexion and extension, performing 4 series of 30/15/15/15 repetitions as usual in this type of interventions.
  Interventions: Other: Muscle strengthening (BFRT)

INTERVENTIONS:
Other: Muscle strengthening (BFRT) — The experimental group will perform a low-intensity strengthening program (20% 1RM) in combination with the BFRT system consisting of the following exercises: palmar flexion and dorsal flexion; ulnar deviation and radial deviation; pronation and supination; elbow flexion and extension, performing 4 sets of 30/15/15/15 repetitions as usual in this type of interventions.
  Once the first exercise has been completed, a rest of 3 - 4 minutes should be taken depending on the fatigue perceived by the patient. Subsequently, the other two exercises will be performed following the scheme already outlined.
  Taking into account the scientific evidence concerning the safety and adverse effects linked to the BFRT system, it is determined that the pressure applied in the experimental protocol will be 60% of the TRP of each subject, following the recommendations that locate the effective pressure between 50 - 80% of the TRP of each subject.
  Arms: BFRT
Other: Conventional physical therapy — The control group will perform a conventional muscle strengthening protocol consisting of the following exercises: palmar flexion and dorsal flexion; ulnar deviation and radial deviation; pronation and supination; elbow flexion and extension, with a dumbbell at 70% of 1RM, performing a total of 4 sets of 8 - 12 repetitions each, avoiding muscle failure in each set.
  Arms: Conventional muscle strengthening

SUMMARY:
Although the Blood Flow Restriction Training (BFRT) system has attracted the attention of health professionals, research on this tool in people with neurological pathology, particularly multiple sclerosis (MS), is very limited. Furthermore, to our knowledge, studies on the effect of the BFRT system on forearm-hand muscle strength and fatigability, coordination and dexterity, functionality and quality of life in people with MS are nonexistent.

The main objective of our study are:

-To know the effects of low intensity training in combination with the BFRT system on upper limb strength and forearm and hand fatigability, dexterity, functionality and quality of life in people with MS.

Secondary Objectives

* To know if a low-intensity muscle strengthening program in combination with the BFRT system is superior to a conventional strengthening program.
* To know the adherence and satisfaction with the experimental intervention.

The investigators propose to conduct a randomized controlled trial (RCT) with examiner blinding with pre-intervention, post-intervention and follow-up assessment, following the recommendations of the CONSORT guidelines, designed to study the effects of the application of a low-intensity muscle strengthening program in combination with the BFRT system. This intervention will be carried out at the Leganés Multiple Sclerosis Association (ALEM). Patients will be randomly assigned through the GraphPad Software® QuickCalcs application to 2 study groups. A control group, which will receive a low intensity strengthening program in combination with the BFRT system; and an experimental group, which will receive a high intensity strengthening program.

Voluntary participation will be requested from patients diagnosed with MS in the Leganés Multiple Sclerosis Association (ALEM) who meet the inclusion criteria. Acceptance of the study and signature of the informed consent form will be required prior to the start of the program.

As this is the first study to evaluate the effectiveness and feasibility of a low-intensity muscle strengthening protocol in combination with BFRT on forearm and hand muscle strength and fatigability, coordination, dexterity, functionality and quality of life in people with MS, the sample size will be determined based on the most similar scientific literature possible. Hill et al developed an investigation comparing the adaptations of MS patients to two types of intervention: high intensity or conventional strengthening program versus low intensity in combination with BFRT. Since this is the only investigation to date that includes MMSS exercises in their intervention, we consider that the sample size proposed by Hill et al is the most appropriate for our investigation. The sample size obtained in that investigation was 19 subjects, so for the sample size of the present investigation a total of 19 subjects is proposed. However, estimating a 10% possible percentage of losses, we estimate a total of 21 total participants to be recruited.

Patients will be randomly assigned via the GraphPad Software® QuickCalcs application to 2 study groups. A control group, which will receive a low-intensity strengthening program in combination with the BFRT system; and an experimental group, which will receive a high-intensity strengthening program.

DETAILED DESCRIPTION:
Among the different physical exercise modalities, Blood Flow Restriction Training (BFRT) appears. This type of approach is a training modality performed with occlusion of blood flow in the extremities, partially restricting arterial flow and venous return of blood to the muscles involved. It is usually, but not always, performed in parallel with LL-RT, with repetitions close to muscle fatigue in each set, however, it can also be performed in parallel with functional or task-focused training, such as horizontal walking, aerobic work on a stationary bike. BFRT is applied via an external pneumatic tourniquet at the proximal end of the upper or lower extremity, applying occlusion pressure that promotes ischemia and blood pooling in the capillary beds of the musculature distal to the tourniquet.

A 2020 investigation by Minitti et al indicated that the physiological mechanism behind the findings in muscle adaptations include acute muscle inflammation, increased recruitment of muscle fibers, decreased myostatins, decreased atrogenesis and satellite cell proliferation. Recent research has highlighted that the processes described above can be evoked in low-load strengthening in combination with the BFRT system, but not through conventional or high-load strengthening. In turn, these benefits have been observed in both young and older adults without increasing muscle damage, inflammation or pain perception.

In the field of physiotherapy, BFRT has gained increasing importance, as it has awakened interest in its application as a complement to therapeutic exercise, especially in those subjects who cannot tolerate high loads due to their clinical considerations. Its validity as a tool has been proven both for sports performance in different populations (elite or amateur athletes; young and older adults with no training experience), and in populations with pathology (older adults with fragility, musculoskeletal rehabilitation, post-surgical or post-immobilization conditions, femoropatellar syndromes, meniscus tears, ligamentous strains, rehabilitation after anterior cruciate ligament surgery, people with type 2 Diabetes Myelitus, people with neurological pathologies, including multiple sclerosis, MS).

The systematic review by Reina-Ruiz et al analyzed the effects of the use of the BFRT system in combination with LL-RT and aerobic exercise in people with different pathologies (anterior cruciate ligament reconstruction, stage two chronic kidney disease, coronary artery disease, end-stage renal disease, elderly comatose patients, knee osteoarthritis and recurrent non-specific low back pain). The results obtained in terms of strength, despite the heterogeneity of the outcome measures used, present the BFRT system as an effective tool for strength improvement, being equal or superior to HL-RT.

In a study conducted in 2022, Vinolo-Gil et al conducted a systematic review on the use of the BFRT system in populations with different neurological pathologies (spinal cord injury (SCI), stroke, cerebral palsy and MS). Their results showed improvements in sensorimotor function, frequency, gait length symmetry, gait speed and muscle thickness. However, no improvements in balance were found. The systematic review by Jønsson et al published in the current year 2024 reported that BFRT generated greater improvements in strength in people with inclusion body myositis compared to those who received no intervention and in subjects with incomplete spinal cord injury who performed the BFRT protocol in combination with functional electrical stimulation (FES), showing greater muscle circumference in the quadriceps than those who only received FES-based treatment, with unclear results in people with MS.

Given the idiosyncrasy of the tool, the safety of its use is a recurring theme in research, so a detailed analysis of the characteristics of the intervention is necessary. Since its origin in the 1980s, different types of cuffs have been used: pneumatic bicycle inner tubes, elastic bands and electronic devices. There is no scientific consensus on the use of one model over another; however, different investigations highlight certain determining characteristics for the safety and efficacy of the tool. The 4 main variables to take into account are: a) restriction pressure; b) cuff width; c) cuff type; d) cuff material.

Another major concern of researchers about the BFRT system is the pain that may result from an intervention with these characteristics, which has increased significantly in recent years in this regard.

The findings in terms of pain should be grouped into 2 sections: short term, medium term and long term. Short term: Korakakis et al analyzed the effects of an exercise protocol based on knee extension with low loads in combination with the BFRT system on anterior knee pain, observing that the 30 intervention subjects reduced their pain level in the 3 tests performed. In turn, the level of analgesia generated was maintained 45 minutes later, after a conventional physiotherapy session. Another investigation by Korakakis et al compared the effects of a low-intensity exercise protocol with a low-intensity exercise protocol in combination with the BFRT system. Analgesia in the low intensity and BFRT group was superior to that of the control group. Twenty percent of the participants in the control group reported greater discomfort after the intervention and 15% after 45 minutes. In turn, Lixandrão et al compared pain levels during and post-exercise compared to conventional training, finding no greater pain in the BFRT group. Medium and long term: Giles et al compared a low-load exercise protocol in combination with the BFRT system versus conventional training in patients with patellofemoral pain. The results showed significant differences in favor of the group that applied the BFRT system; in turn, the improvements were maintained in the follow-up assessment 6 months later.

Beyond pain, the potential adverse effects derived from the BFRT system have been investigated in different investigations, finding no adverse effects in people with neurological pathology according to the systematic review by Jønsson et al of 2024 or only minor adverse effects in populations without neurological pathology such as small hematomas, paresthesias, stiffness, pain or stiffness. According to Nakajima et al (50), from a population of 13,000 subjects without neurological pathology, serious adverse effects derived from an intervention through the BFRT system were extremely rare (0.008-0.055%), some of these being rhabdomyolysis or thromboembolism. With respect to serious adverse effects, it should be noted that the research by Minniti et al (22) presented similar findings in terms of the frequency of occurrence of adverse effects, however, they include an analysis of the cases that presented such serious adverse effects. One patient presented deep vein thrombosis (DVT) having been exposed to continuous occlusion for 30 - 60 minutes and presenting a history of edema and alterations of sensibility of several years of evolution. Two subjects presented rhabdomyolysis, the first had a history of DVT after ankle surgery and was exposed to an arbitrary compression of 100mmHg; the second patient showed no history or apparent risk factors, but the investigators do not know the information regarding the pressure applied and the duration of this. Finally, it is worth noting that in the first case, once he was medicated for the rhabdomyolysis and the patient continued with the experimental protocol without any other adverse effects.

Although the BFRT system has attracted the attention of health professionals, research on this tool in people with neurological pathology, particularly MS, is very limited. Furthermore, to our knowledge, studies on the effect of the BFRT system on forearm-hand muscle strength and fatigability, coordination and dexterity, functionality and quality of life in people with MS are nonexistent.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age.
* Diagnosis of MS according to McDonald criteria (53) with a time of evolution longer than two years.
* Assessment on the Kurtzke Multiple Sclerosis Disability Status Scale (EDSS) with a score between 2. 0 (minimal disability in one section of the FS (at least one with a score of 2).) to 7.0 (unable to walk more than a few steps, even with assistance, basically confined to wheelchair and able to transfer from wheelchair to another place, or can manage to go to the toilet for 12 hours a day) .
* Stable medical treatment for at least six months prior to surgery.
* Upper extremity muscle tone no greater than 2 points (moderate hypertonia, increased muscle tone during most of the arc of motion, but can passively move the affected part with ease) on the modified Ashworth Scale.
* Muscle balance equal to or greater than 3 in the upper extremity.
* Score less than or equal to 4 points on the "Pyramidal Function" section of the EDSS functional scale.
* Absence of cognitive impairment, with ability to understand instructions and score equal to or greater than 24 on the Minimental Test.
* A score equal to or less than 2 points on the "Mental Functions" section of the EDSS.

Exclusion Criteria:

* Diagnosis of a neurological disease or musculoskeletal disorder other than MS.
* Diagnosis of a cardiovascular, respiratory or metabolic disease or other conditions that may interfere with this study.
* Having suffered an exacerbation or hospitalization in the last 3 months before starting the assessment protocol, or during the therapeutic intervention process.
* Having received a course of steroids, intravenous or oral, 6 months prior to the start of the assessment protocol and within the intervention period of the study duration.
* Having received treatment with botulinum toxin in the 6 months prior to the start of the study.
* A score higher than 2 points on the modified Ashworth scale.
* Cognitive or language impairment that prevents adequate communication or comprehension.
* Medical complications such as: history of deep vein thrombosis, pulmonary embolism, vascular disease, thrombophilia, or any circulatory or coagulation disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Isometric prehensile hand strength (Kg) | Up to 8 weeks
  Isometric prehensile hand strength: measured by the JAMAR® fist dynamometer. The JAMAR® dynamometer has been widely cited and is considered the gold standard for the assessment of fist strength. Three measurements of the maximum voluntary maximum isometric contraction (MVC) will be taken with each hand, always starting with the least affected hand; once the three measurements have been taken, the mean of these will be obtained.
  Major values (Kg) means a higher hand grip strengh (there is not a maximum).

SECONDARY OUTCOMES:
Isometric pincer force (Kg) | Up to 8 weeks
  Isometric pincer force: a Baseline Pinch Gauge® will be used to assess 3 different types of pinch: terminal opposition grip, in which the anterior and distal face of the first finger contacts the anterior face of the dynamometer, anterior and distal face of the second finger contacts the posterior face of the dynamometer; pulpolateral grip, in which the anterior face of the distal phalanx of the first finger contacts the anterior face of the dynamometer, radial edge of the second finger contacts the posterior face of the dynamometer; tridigital press of the first three fingers, in which the anterior and distal face of the first finger contacts the posterior face of the dynamometer, anterior and distal face of the second and third finger contacts the anterior face of the dynamometer. As in the previous test, 3 measurements will be taken and the average score will be obtained.
  Major values (Kg) means a better pincer force strengh (there is not a maximum)
Gross coordination for the upper limb (Block and Box; number of cubes) | Up to 8 weeks
  Box and Block Test (BBT): it will be used to assess coordination and manual dexterity. The patient is seated with the tool, a wooden box divided into two identical halves inside which there are 150 wooden cubes of 2.5 cm of different colors, in front of his midline. The patient has to move as many cubes as possible from one half of the box to the other in 60 seconds. The test is performed first with the dominant hand and then with the non-dominant hand. It is a standardized tool for the measurement of the gross function of the MMSS, having been validated by gender and age in healthy subjects, in turn, it shows a low ceiling and floor effect in people with MS.
  pincer force A higher number of cubes (there is not a maximun) indicate a better coordination of the upper limb.
Fine coordination for the upper limb (NHPT; time in seconds) | Up to 8 weeks
  Nine Hole Peg Test (NHPT): this test will be used to assess the function of the MMSS, in particular the fine motor skills of the hand. The tool will be placed in front of the subject's midline, the subject will have to insert the 9 pegs, one at a time, into the 9 holes of a board and then remove them, again one at a time, in the shortest possible time; first with the dominant hand, and then the non-dominant hand, the hand that is not being assessed can hold the board to provide stability. The score is the time in seconds required to insert and remove all the pins. It shows excellent test-retest, inter-rater and inter-rater reliability and adequate internal consistency.
  Lower time in seconds (s) (not specificated the minimum) in the test indicates a better fine coordination.
Functional status of the upper limb (ABILHAND) | Up to 8 weeks
  Abilhand: is a self-administered questionnaire to assess the person's manual dexterity, defining this as the ability to perform a series of tasks, regardless of the strategies applied to achieve it. The questionnaire contains 23 items scored from 0 to 2, which correspond to various ADL tasks; the patient will mark the degree of difficulty he or she refers to when performing the activities. The score can range from 0 to 46 points, the higher the score, the better the manual dexterity. Its inter- and intra-rater reliability, internal consistency and construct validity are excellent.
  A higher score (maximun 46 points) indicates a better functionality.
Quality of life (MSIS-29) | Up to 8 weeks
  Multiple Sclerosis Impact Scale (MSIS-29): is a self-applied scale on the impact of the disease on the patient's life in the two weeks prior to performing. It presents 29 questions of which 20 assess the physical aspects of MS and 9 assess the psychosocial aspects. The physical sphere has been proven to have high internal consistency and good construct validity, while the cognitive sphere has good internal consistency.
  A higher score (maximun 29 points) indicates a better quality of life.
Satisfaction (CSQ8) | Up to 8 weeks
  CSQ8: self-completed questionnaire with eight dimensions measuring satisfaction with the care and treatment received. The total score is 32 points, where maximum scores indicate higher satisfaction. Dimensions related to satisfaction with the training modality and tool used (entertainment, ease of use, accessibility, among others), the professional who applies it (clear explanation, availability, adaptability, among others) or recommendation to other patients will be evaluated.
  A higher score (maximun 32 points) indicates a better satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Cano de la Cuerda, PT, PhD, Principal Investigator — Universidad Rey Juan Carlos
Locations (1):
- Universidad Rey Juan Carlos, Alcorcón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No